CLINICAL TRIAL: NCT05622682
Title: A Prospective Cohort Study to Define Infectious Burden, the Seroprevalence of Vaccine Preventable Pathogens and Immune Recovery in the First Year Following Completion of Therapy in Patients With Acute Lymphoblastic Leukemia (ALL)
Brief Title: Vaccine Immune Recovery After Leukemia
Acronym: VIRAL
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-019426; 61366 (Other Grant/Funding Number: Merck Sharp and Dohme LLC)
Record Dates: First submitted 2022-11-09; First posted 2022-11-18 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
Keywords: acute lymphoblastic leukemia; chemotherapy; antineoplastic agents; varicella vaccine; chickenpox vaccine; pneumococcal vaccines; measles vaccine
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children, adolescents, and young adults who recently completed ALL treatment: This cohort of participants who recently completed leukemia therapy will be assessed for infection incidence during the year following treatment and give blood samples to be measured for antibodies to vaccine-preventable diseases. A small subset will also have their blood samples tested for B and T cell recovery.
  Interventions: Other: Observational only: Serology and flow cytometry for ALL cohort participants; Other: Observational only: Infection rates

INTERVENTIONS:
Other: Observational only: Serology and flow cytometry for ALL cohort participants — Blood samples from ALL cohort participants will be tested to measure antibodies to vaccine-preventable diseases and immune recovery
Other: Observational only: Infection rates — Number of infections during the study period will be obtained and infection incidence rates calculated during the first year off-chemotherapy.

SUMMARY:
This observational study aims to assess recovery of the immune system and immunity to vaccine-preventable diseases in children, adolescents, and young adults who recently completed treatment for acute lymphoblastic leukemia (ALL). Several children's hospitals in the United States are participating in the study, which will enroll up to 100 pediatric participants. The study is intended to determine the rate of infection after leukemia treatment and to inform future studies and recommendations about whether children and adolescents who have leukemia should receive additional vaccine doses or boosters after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents, and young adults diagnosed with B or T ALL at age 12 months or older
* Completed ALL chemotherapy within the past three months or will complete ALL chemotherapy in the upcoming three months
* Three years of age or older at time of enrollment

Exclusion Criteria:

* Diagnosis of infant ALL
* Evidence of disease relapse
* History of primary immunodeficiency (except related to Down Syndrome)
* History of a stem cell transplant or cellular immunotherapy
* History of prior malignancy or condition requiring chemotherapy other than for current ALL diagnosis

Ages: 3 Years to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, adolescents, and young adults receiving care at a participating pediatric oncology/hematology center who recently completed or will soon complete treatment for acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian T Fisher, DO MSCE MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (6):
- United States (6):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - CHRISTUS Children's (Affiliate of Baylor College of Medicine), San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: September 2022 - October 2024 Participating sites: Six pediatric hemotology/oncology centers in the U.S. Patients completing chemotherapy for acute lymphoblastic leukemia during the study period screened for eligibility.
Pre-assignment Details: This was an observational study with only one study arm for enrollment of participants recently completing chemotherapy for acute lymphoblastic leukemia.
Groups:
- Child, Adolescent, and Young Adult Survivors of Acute Lymphoblastic Leukemia: This group includes survivors of acute lymphoblastic leukemia between ages 3 and 31 who completed chemotherapy for acute lymphoblastic leukemia within +/- 3 months of the time of study enrollment and were followed until one year off-therapy.
Period: Overall Study
Arm/Group | Child, Adolescent, and Young Adult Survivors of Acute Lymphoblastic Leukemia
Started | 89
3 Months Off-therapy Follow-up | 88
6 Months Off-therapy Follow-Up | 86
12 Months Off-therapy Follow-up | 84
Completed | 84
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Censored Due to ALL Relapse | 3

BASELINE CHARACTERISTICS:
Arm/Group | Child, Adolescent, and Young Adult Survivors of Acute Lymphoblastic Leukemia
Number analyzed (Participants) | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 57
  More than one race | 3
  Unknown or Not Reported | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 78
  Unknown or Not Reported | 0
Acute Lymphoblastic Leukemia Subtype and Risk Classification [Count of Participants; unit: Participants]
  Standard-risk B-cell Acute Lymphoblastic Leukemia | 47
  High-risk B-cell Acute Lymphoblastic Leukemia | 27
  T-cell Acute Lymphoblastic Leukemia | 15
Age, Continuous [Median (Inter-Quartile Range); unit: Years] — Age at Study Enrollment in Years
  Years | 8.7 [5.6 to 12.7]
Age, Continuous [Median (Inter-Quartile Range); unit: Years] — Age at Diagnosis of Acute Lymphoblastic Leukemia in Years Population: Age at which study participants were first diagnosed with acute lymphoblastic leukemia.
  Years | 6.0 [3.0 to 10.2]

OUTCOME MEASURES:

1. Primary Outcome: Incident Infection Rate in Participants During the First Year Post-acute Lymphoblastic Leukemia Therapy
Description: Infections include clinical and/or microbiologically confirmed infections as well as patient-reported infections during follow-up. All unique infections for a given subject will be captured and included in the final infection rate per person time estimate. The total number of unique infections identified within the first year after completing chemotherapy will be reported as a rate per patient-year. Patients will be censored at time of loss to follow-up, relapse, or death.
Time Frame: 1 year
Population: Analyzed 88 total participants; 1 participant lost to follow-up between enrollment and first post-enrollment study encounter.
Measure: Number; unit: Events per person-year
Arm/Group | Child, Adolescent, and Young Adult Survivors of Acute Lymphoblastic Leukemia
Number analyzed (Participants) | 88
Events per person-year | 3.60

2. Secondary Outcome: Proportion of Patients With Seroprevalence of Measles Antibodies at Each Study Timepoint
Description: The seroprevalence proportions for measles antibodies will be determined for the entire cohort and by demographics at each study follow-up time point (3, 6, and 12 months). Additionally, seroprevalence at each time point will be described for participants who had and had not completed their primary vaccine series before starting chemotherapy.
Time Frame: 1 year
Population: For each timepoint, only patients with (A) any history of measles vaccine prior to chemotherapy and NO history of measles vaccine after chemotherapy and (B) serum available for testing at the timepoint are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Child, Adolescent, and Young Adult Survivors of Acute Lymphoblastic Leukemia
Number analyzed (Participants) | 88
Participants
  Measles-specific Immunoglobulin-G Level Indicative of Seroprotection at 3 Months Off-therapy: number analyzed (Participants) | 58
  Measles-specific Immunoglobulin-G Level Indicative of Seroprotection at 3 Months Off-therapy | 37
  Measles-specific Immunoglobulin-G Level Indicative of Seroprotection at 6 Months Off-therapy: number analyzed (Participants) | 60
  Measles-specific Immunoglobulin-G Level Indicative of Seroprotection at 6 Months Off-therapy | 30
  Measles-specific Immunoglobulin-G Level Indicative of Seroprotection at 12 Months Off-therapy: number analyzed (Participants) | 64
  Measles-specific Immunoglobulin-G Level Indicative of Seroprotection at 12 Months Off-therapy | 29

3. Secondary Outcome: Proportion of Patients With Seroprevalence of Varicella Antibodies at Each Study Timepoint
Description: The seroprevalence proportions for varicella antibodies will be determined for the entire cohort and by demographics at each study follow-up time point (3, 6, and 12 months). Additionally, seroprevalence at each time point will be described for participants who had and had not completed their primary vaccine series before starting chemotherapy.
Time Frame: 1 year
Population: For each timepoint, participants with (A) any history of varicella vaccine prior to chemotherapy and NO history of varicella vaccine after chemotherapy and (B) serum available for testing at the timepoint are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Child, Adolescent, and Young Adult Survivors of Acute Lymphoblastic Leukemia
Number analyzed (Participants) | 88
Participants
  Varicella-specific Immunoglobulin-G Level Indicative of Seroprotection at 3 Months Off-therapy: number analyzed (Participants) | 58
  Varicella-specific Immunoglobulin-G Level Indicative of Seroprotection at 3 Months Off-therapy | 9
  Varicella-specific Immunoglobulin-G Level Indicative of Seroprotection at 6 Months Off-therapy: number analyzed (Participants) | 61
  Varicella-specific Immunoglobulin-G Level Indicative of Seroprotection at 6 Months Off-therapy | 8
  Varicella-specific Immunoglobulin-G Level Indicative of Seroprotection at 12 Months Off-therapy: number analyzed (Participants) | 65
  Varicella-specific Immunoglobulin-G Level Indicative of Seroprotection at 12 Months Off-therapy | 11

4. Secondary Outcome: Proportion of Patients With Seroprevalence of Pneumococcus Antibodies at Each Study Timepoint
Description: The seroprevalence proportions for pneumococcal antibodies (23 serotypes) will be determined for the entire cohort and by demographics at each study follow-up time point (3, 6, and 12 months). Additionally, seroprevalence at each time point will be described for participants who had and had not completed their primary vaccine series before starting chemotherapy.
Time Frame: 1 year
Population: Patients with any history of pneumococcal vaccine and serum available for testing at each timepoint were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Child, Adolescent, and Young Adult Survivors of Acute Lymphoblastic Leukemia
Number analyzed (Participants) | 79
Participants
  Patients with Positive Titers to > 50% of Pneumococcal Vaccine Serotypes at 3 Months Off-therapy: number analyzed (Participants) | 72
  Patients with Positive Titers to > 50% of Pneumococcal Vaccine Serotypes at 3 Months Off-therapy: Positive Titers Among Patients with Pneumococcal Vaccine Only Pre-chemo | 0
  Patients with Positive Titers to > 50% of Pneumococcal Vaccine Serotypes at 3 Months Off-therapy: Positive Titers Among Patients with Vaccine Pre-chemo and Post-chemo Booster | 0
  Patients with Positive Titers to > 50% of Pneumococcal Vaccine Serotypes at 3 Months Off-therapy: Negative Titers | 72
  Patients with Positive Titers to > 50% of Pneumococcal Vaccine Serotypes at 6 Months Off-therapy: number analyzed (Participants) | 75
  Patients with Positive Titers to > 50% of Pneumococcal Vaccine Serotypes at 6 Months Off-therapy: Positive Titers Among Patients with Pneumococcal Vaccine Only Pre-chemo | 0
  Patients with Positive Titers to > 50% of Pneumococcal Vaccine Serotypes at 6 Months Off-therapy: Positive Titers Among Patients with Vaccine Pre-chemo and Post-chemo Booster | 1
  Patients with Positive Titers to > 50% of Pneumococcal Vaccine Serotypes at 6 Months Off-therapy: Negative Titers | 74
  Patients with Positive Titers to > 50% of Pneumococcal Vaccine Serotypes at 12 Months Off-therapy: Positive Titers Among Patients with Pneumococcal Vaccine Only Pre-chemo | 4
  Patients with Positive Titers to > 50% of Pneumococcal Vaccine Serotypes at 12 Months Off-therapy: Positive Titers Among Patients with Vaccine Pre-chemo and Post-chemo Booster | 4
  Patients with Positive Titers to > 50% of Pneumococcal Vaccine Serotypes at 12 Months Off-therapy: Negative Titers | 71

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow up, approximately 1 year
Description: This study was observational in nature. Participants were monitored for death, relapse of acute lymphoblastic leukemia, or diagnosis of secondary malignancy during the follow-up period.
Arm/Group | Child, Adolescent, and Young Adult Survivors of Acute Lymphoblastic Leukemia
All-Cause Mortality (participants affected / at risk) | 0/89
Serious Adverse Events (participants affected / at risk) | 3/89
Other Adverse Events (participants affected / at risk) | 0/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Child, Adolescent, and Young Adult Survivors of Acute Lymphoblastic Leukemia (N=89)
Relapse of acute lymphoblastic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 — Participants were monitored for relapse of acute lymphoblastic leukemia and censored at the time of relapse diagnosis.
Diagnosis of secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0

LIMITATIONS AND CAVEATS:
This study has several limitations. Because research blood draws were timed with clinical laboratory draws at off-therapy visits, only patients with consistent follow-up were included in the vaccine titer data. Similarly, for infection incidence rates, only patients who consistently followed up and participated in study encounters were captured, meaning that some infections - perhaps among patients more likely to be ill - may have been missed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT05622682/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT05622682/ICF_001.pdf